CLINICAL TRIAL: NCT00801320
Title: Study of Primary Tumor Harvest for the Purpose of Possible Use in a Future Clinical Trial in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Cancer (Ovarian Spore)
Brief Title: Primary Tumor Harvest for the Purpose of Possible Use in a Future Clinical Trial in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Avigan, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 07-319
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: tumor harvest; tumor collection; tumor storage
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Patients with either primary ovarian carcinoma or ovarian carcinoma in first relapse treated with DC/Ovarian tumor cells + GM-CSF
  Interventions: Procedure: Tumor collection
- Cohort 2 (Experimental): Patients with either primary ovarian carcinoma or ovarian carcinoma in first relapse treated with DC/Ovarian tumor cells + GM-CSF and topical Imiquimod at site of vaccination
  Interventions: Procedure: Tumor collection

INTERVENTIONS:
Procedure: Tumor collection — Tumor collected at the time of planned surgery

SUMMARY:
The purpose of this research study is to collect tumor samples at the time of surgery and store them for possible use as part of an experimental vaccine study for the participants cancer in the future.

DETAILED DESCRIPTION:
* Even if tumor sample is collected, the participant is under no obligation to participate in the vaccine study.
* Participants will have their regularly planned surgery as described by their surgeon. During the surgery, tumor samples will be collected. We will only collect tumor that is not needed and could otherwise be thrown away.
* The tumor samples will be frozen and placed in storage for up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of advanced ovarian, fallopian tube or primary peritoneal cancer as determined by a gynecologic oncologist
* Patients are planning to undergo primary or secondary debulking surgery as part of standard of care for their disease
* Estimated life expectancy of 6 months or greater
* 18 years of age or older

Exclusion Criteria:

* More than one prior chemotherapy regimen
* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, unstable ischemic coronary disease or congestive heart failure
* Known HIV infection
* Active second malignancy, aside from basal cell or squamous cell carcinoma of the skin
* Significant autoimmune disease, including psoriasis
* History of clinically significant venous thromboembolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
To collect patient tumor samples that could possibly be used in a subsequent clinical vaccine trial (DF/HCC protocol 07-380). | 2 years
To gain experience in appropriate clinical processing of tumor samples and determining cell yield. | 2 years

SECONDARY OUTCOMES:
Based on feasibility of collection of blood samples of subjects, quantification of T cell subsets, regulatory T cells, activated memory effector cells, and DC phenotype at pre-surgery and post-surgery time points. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts